CLINICAL TRIAL: NCT03439891
Title: Multicenter Pilot Study of the Safety, Efficacy, and Immune Cell Profiling in Advanced Hepatocellular Carcinoma (HCC) Patients Treated With the Combination of Sorafenib Plus Nivolumab as First-Line of Systemic Therapy
Brief Title: Sorafenib and Nivolumab in Treating Participants With Unresectable, Locally Advanced or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robin Kate Kelley (Other)
Collaborators: Bayer (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Robin Kate Kelley, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 174523; NCI-2018-00051 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v7; Stage IIIC Hepatocellular Carcinoma AJCC v7; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: Starting Dose Schedule (DL -1) Once a day (Experimental): Participants with Child-Pugh A or B7 receive a daily dose of 400mg sorafenib on days 1-28, and 240mg of nivolumab IV over 30 minutes beginning on day 15 of course 1, then on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course will continue until 1 dose-limiting toxicity occurs to establish maximum tolerated dosing schedule.
  Interventions: Biological: Nivolumab; Drug: Sorafenib
- Part 1: Escalated Dose Schedule (DL 1) Twice a day (Experimental): Participants with Child-Pugh A or B7 receive a daily dose of 400mg sorafenib twice a day on days 1-28, and 240mg of nivolumab IV over 30 minutes beginning on day 15 of course 1, then on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course will continue until 1 dose-limiting toxicity occurs to establish maximum tolerated dosing schedule.
  Interventions: Biological: Nivolumab; Drug: Sorafenib
- Part 2: Child-Pugh B (CPB) Expansion Cohort (sorafenib, nivolumab) (Experimental): Participants with Child-Pugh B7-9 receive sorafenib at the maximum tolerated dose (MTD) established in Part 1 on days 1-28, and nivolumab IV over 30 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Drug: Sorafenib

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Sorafenib — Given PO
  Other Names: BAY 43-9006

SUMMARY:
This phase II trial studies the best dose and side effects of sorafenib tosylate and nivolumab in treating patients with liver cancer that cannot be removed by surgery (unresectable), has spread to nearby tissues or lymph nodes (locally advanced) or to other places in the body (metastatic). Sorafenib tosylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving sorafenib tosylate and nivolumab may work better in treating patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Maximum tolerated dose (MTD) of sorafenib tosylate (sorafenib) in combination with standard dose nivolumab with Child Pugh A-B7 liver function. (Part 1: Escalation Cohort).

II. Safety in participants with Child-Pugh B liver function. (Part 2: Child-Pugh B Escalation Cohort)

SECONDARY OBJECTIVES:

I. Safety and tolerability of combination overall. (Parts 1 and 2).

II. Rate of immune-related adverse event (irAE) for combination overall and in participants with Child-Pugh B liver function. (Parts 1 and 2).

III. Overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in participants with Child-Pugh B liver function. (Parts 1 and 2).

IV. Duration of response (DOR), progression free survival (PFS), and overall survival (OS) for escalation cohort and Child-Pugh B expansion cohort and overall. (Parts 1 and 2).

EXPLORATORY OBJECTIVES:

I. Relationship between peripheral blood mononuclear cell (PBMC) immune cell subset frequencies, baseline liver function, and clinical outcomes.

II. Relationship between PBMC T cell receptor (TCR) clonotype frequency and diversity, baseline liver function, and clinical outcomes.

III. Tumor tissue immune cell subsets and TCR clonotype frequency and diversity in pre-treatment archival tumor tissue samples.

IV. Tumor and immune cell programmed death-ligand 1 (PD-L1) status in pre-treatment archival tumor tissue samples and relationship to clinical outcomes.

V. Changes in hepatitis B virus (HBV) and/or hepatitis C virus (HCV) viral load on treatment.

VI. Alpha-fetoprotein (AFP) changes on treatment and relationship to clinical outcomes.

VII. Relationship between clinical outcomes and clinicopathologic features including race/ethnicity, etiology of liver disease including HBV/HCV status, baseline liver function, presence of cirrhosis, macrovessel invasion, extrahepatic spread, site(s) of metastatic disease, prior treatment history including prior radiation and arterial therapies.

OUTLINE: This is a dose-escalation and expansion study of sorafenib tosylate.

DOSE-ESCALATION (Part 1):

Between 3-12 participants will be enrolled in Part 1. Participants receive sorafenib tosylate orally (PO) once daily (QD) or twice daily (BID) on days 1-28, and nivolumab intravenously (IV) over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

EXPANSION COHORT (Part 2).

Participants receive nivolumab IV over 30 minutes on days 1 and 15, and sorafenib tosylate once daily (QD) or twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 and 100 days, then every 3 months for up to 2 years after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of unresectable, locally advanced and/or metastatic hepatocellular carcinoma (HCC) not amenable to curative surgery, transplantation, or ablative therapies based upon assessment of treating investigator.

   a. For patients without prior histologic or cytologic diagnosis, radiographic diagnosis is allowed provided patients meet American Association for the Study of Liver Diseases (AASLD) criteria for radiographic diagnosis.
2. Radiographically measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 in at least one site not previously treated with chemoembolization, radioembolization, radiation, or other local/liver-directed procedures (i.e. must have at least one measurable target lesion, either within the liver or in a measurable metastatic site); a new area of tumor progression within or adjacent to a previously-treated lesion, if clearly measurable by a radiologist, is acceptable.
3. Untreated/pretreatment archival tumor tissue must be available for correlative analyses
4. Age at least 18 years at enrollment.
5. Eastern Cooperative Oncology Group (ECOG) 0 or 1 at enrollment
6. At least 4 weeks after any prior chemoembolization, radioembolization, local ablative therapies, or hepatic radiation and recovery to =< grade 1 treatment-related toxicity.
7. At least 6 weeks after any major surgery including prior hepatic resection and recovery to =< grade 1 treatment-related toxicity.
8. At least 7 days after minor surgery (such as central venous access) or biopsy and recovery to =< grade 1 treatment-related toxicity
9. At least 2 weeks after any prior palliative radiation (e.g. to focal metastatic lesion such as bone metastases) and recovery to =< grade 1 treatment-related toxicity.
10. Blood pressure =< 140/90 mm Hg with or without anti-hypertensive therapy

    a. Patients may be rescreened after initial ineligibility if due to elevated blood pressure, if adequately medically managed within approximately 30 days.
11. Adequate baseline organ and marrow function as defined below:

    1. Adequate bone marrow function:

       * Absolute neutrophil count at least 1,200/microliter (mcL).
       * Platelets at least 50,000/mcL.
       * Hemoglobin at least 9 g/dL.
    2. Adequate hepatic function:

       * Part 1: Total bilirubin less than 2.6 mg/dL or 2 times upper limit of normal (ULN), whichever is higher, and albumin at least 2.5 g/dL, if otherwise meets criteria for Child Pugh A or B7.
       * Part 2: Total bilirubin less than 3.9 mg/dL or 3 times ULN, whichever is higher, and albumin at least 2.0 g/dL, if otherwise meets criteria for Child Pugh B.
       * Both Parts: Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) less than 5 X ULN, International normalized ratio (INR) less than 1.7.
    3. Creatinine less than 1. 5 X ULN and/or creatinine clearance >= 60 mL/min.
12. Child-Pugh A or B7 (Part 1); Child-Pugh B7-9 (Part 2).
13. If HBV surface antigen (sAg) and/or core antibody (Ab) positive, must be treated with appropriate antiviral therapy according to institutional practice with HBV deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR) less than 500 IU/mL.
14. If clinical or histologic diagnosis of cirrhosis and/or clinical or radiographic evidence esophageal or gastric varices, must have had esophagogastroduodenoscopy (EGD) surveillance and adequate endoscopic therapy according to institutional standards.
15. Able to swallow and retain oral medications
16. Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 28 days before study enrollment.
17. WOCBP and male partners of WOCBP must agree to use two methods of contraception until at least 5 months after last dose of each study drug for WOCBP subjects, and 7 months for male partners of WOCBP.
18. Able to understand and willingness to provide informed consent, and the willingness to comply with the requirements of the protocol.

    1. Subjects must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committees (IEC) approved written informed consent form in accordance with regulatory and institutional guidelines and before the performance of any protocol related procedures that are not part of standard of care.

Exclusion Criteria:

1. Any prior systemic therapy for HCC.
2. Known fibrolamellar or mixed HCC-cholangiocarcinoma histology.
3. Requirement for paracentesis to control ascites within 6 months before enrollment.

   a. Ascites which is not clinically detectable or mild on stable doses of diuretics during screening is allowed provided meets criteria for Child Pugh A or B7 (Part 1) or B7-9 (Part 2).
4. Symptomatic hepatic encephalopathy requiring medication (such as lactulose or rifaximin) (Part 1) or any hospitalization for encephalopathy within 6 months before enrollment (Part 1 or 2).

   1. Hepatic encephalopathy that is adequately controlled on stable doses of lactulose and/or rifaximin per assessment of treating investigator is allowed in Part 2, provided no hospitalization for encephalopathy within 6 months before enrollment.
   2. Medications such as lactulose used for other indications (e.g. constipation) are allowed in both Part 1 and 2.
5. History of upper gastrointestinal (GI) bleeding from esophageal and/or gastric varices within 12 months before enrollment.
6. Requirement for systemic corticosteroids unless used for adrenal replacement, acute therapy for asthma or bronchitis exacerbation (=< 2 weeks), or premedication for contrast allergy.

   a. Topical, intranasal, or inhaled steroids are not excluded.
7. Active autoimmune condition requiring systemic immunosuppressive medication.
8. Known human immunodeficiency virus (HIV) infection.
9. Active coinfection with HBV plus hepatitis delta (D) virus (HDV) or HCV:

   1. Both hepatitis B and C as evidenced by detectable HBV surface antigen or HBV DNA and detectable HCV ribonucleic acid (RNA).
   2. Hepatitis D infection (HDV antibody positive) in subjects with detectable hepatitis B surface antigen or HBV DNA.
10. Prior allogeneic transplant of any solid organ or bone marrow/stem cells.
11. Symptomatic hypothyroidism without replacement.

    a. Patients may be rescreened after initiating adequate replacement therapy
12. History of seizure disorder requiring antiepileptic medication or brain metastases with seizures.
13. Non-healing wound, ulcer, non-healing traumatic bone fracture, or abscess within 30 days of enrollment.

    a. Nondisplaced, uncomplicated pathologic fracture due to tumor may be eligible provided adequately treated with radiation, surgery or other treatments with full recovery based upon investigator assessment.
14. Central or necrotic lung metastases.
15. Known brain or leptomeningeal metastases.
16. Uncontrolled hypertension (systolic pressure > 140 mm Hg and/or diastolic pressure > 90 mm Hg (National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v4.0) on repeated measurement) despite optimal medical management.
17. Active or clinically significant cardiac disease including:

    1. Congestive heart failure - New York Heart Association (NYHA) > class II.
    2. Active coronary artery disease including unstable or newly diagnosed angina or myocardial infarction within 6 months prior to study entry.
    3. Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
    4. Corrected QT interval (QTc) (Fridericia) > 450 msec on two consecutive electrocardiograms (ECGs) (baseline ECG should be repeated if QTc is found to be > 450 msec).
18. Subject with any pulmonary hemorrhage/bleeding event of NCI-CTCAE v4.0 grade 2 or higher within 6 months before first dose of study treatment any other hemorrhage/bleeding event of NCI-CTCAE v4.0 grade 3 or higher within 6 months before first dose of study treatment.
19. Subjects with arterial or venous thrombotic or embolic, such as cerebrovascular accident (including transient ischemic attacks), myocardial infarction, or deep venous thrombosis (DVT) within 6 months of informed consent.

    1. Tumor or bland thrombus in hepatic vasculature is not an exclusion provided hepatic function criteria are met.
    2. Asymptomatic thromboembolic events such as incidentally-detected sub-segmental pulmonary emboli or superficial thromboses are not an exclusion provided the patient does not require treatment with therapeutic anticoagulation.
20. Subjects who have used strong CYP3A4 inducers (eg, phenytoin, carbamazepine, phenobarbital, St. John's wort (hypericum perforatum), dexamethasone at a dose of greater than 16 mg daily, or rifampin [rifampicin], and/or rifabutin) within 28 days before first dose of study treatment.
21. Subjects who require therapeutic anticoagulation or anti-platelet therapy.

    1. Low dose aspirin (=< 100 mg/day) is allowed
    2. Prophylactic doses of low molecular weight heparin (LMWH) are allowed if approved by study chair or designee.
22. Subjects with any previously untreated and concurrent cancer that is distinct in primary site or histology from HCC except cervical cancer in-situ, treated nonmelanoma skin cancers, localized prostate cancer not requiring systemic therapy undergoing surveillance, or superficial bladder tumor; subjects surviving a cancer that was curatively treated and without evidence of disease for more than 2 years before enrollment are allowed provided that cancer therapy was completed at least 2 years prior to study entry (date of the informed consent form).
23. Any uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring antibiotic therapy, pulmonary disease impairing functional status or requiring oxygen, impairment in gastrointestinal function that may affect or alter absorption of oral medications (such as malabsorption or history of gastrectomy or bowel resection), or uncontrolled diarrhea.
24. Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
25. Women who are pregnant or breast-feeding at enrollment
26. Inability to comply with the protocol and/or not willing or not available for follow-up assessments.
27. Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin K. Kelley, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The intent of the addition of Part 2 for Child-Pugh B participants in the protocol was to capture the differences in treatment outcomes for those with Child-Pugh A (CPA) versus Child-Pugh B (CPB). The single participant with CPB enrolled to Part 1 of the study was therefore included in some of the efficacy analyses focused on outcomes for CPB participants specifically.
Groups:
- Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab): Participants with Child-Pugh B7-9 receive sorafenib at the MTD established in Part 1 on days 1-28, and nivolumab IV over 30 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Study Cohort Assignment
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab)
Started | 6 | 5 | 5
Completed | 6 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Parts 1 & 2: All CPB Participants
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab)
Started | 0 | 1 | 5
Completed | 0 | 1 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Starting Dose Schedule (DL -1) Once a Day: Participants with Child-Pugh A - B7 receive a daily dose of 400mg sorafenib on days 1-28, and 240mg of nivolumab IV over 30 minutes beginning on day 15 of course 1, then on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course will continue until 1 dose-limiting toxicity occurs to establish maximum tolerated dosing schedule.
- Part 1: Escalated Dose Schedule (DL 1) Twice a Day: Participants with Child-Pugh A - B7 receive a daily dose of 400mg sorafenib twice a day on days 1-28, and 240mg of nivolumab IV over 30 minutes beginning on day 15 of course 1, then on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course will continue until 1 dose-limiting toxicity occurs to establish maximum tolerated dosing schedule.
- Part 2: Child Pugh B Expansion (Sorafenib, Nivolumab): Participants with Child-Pugh B7-9 receive sorafenib at the MTD established in Part 1 on days 1-28, and nivolumab IV over 30 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion (Sorafenib, Nivolumab) | Total
Number analyzed (Participants) | 6 | 5 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (4.5) | 66 (11.4) | 67 (6.6) | 65.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 5 | 3 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 4 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 3 | 1 | 4 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 5 | 16
Child-Pugh Classification and Score [Count of Participants; unit: Participants] — The Child-Pugh classification is a system for assessing the prognosis of chronic liver disease, primarily cirrhosis and determined by scoring clinical measures of liver disease and possibility of eventual liver failure. Each person is assigned a classification and score summarizing the prognosis: Class A (5-6 points, least severe liver disease, one to five-year survival rate: 95 percent), Class B (7-9 points, moderately severe liver disease one to five-year survival rate: 75 percent) or Class C (10-15 points most severe liver disease one- to five-year survival rate: 50 percent).
  Participants
    Child-Pugh A | 6 | 4 | 0 | 10
    Child-Pugh B | 0 | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Part 1 Only)
Description: MTD is defined as the dose in which 1 or more dose limiting toxicities (DLT) is reported by study participants in Part 1 within the first cycle of treatment. Participants in Part 1 must receive at least 2 doses of nivolumab and at least 75% of sorafenib doses within 28 days (1 cycle), or experience a qualifying DLT event to be evaluable.
Time Frame: 28 days
Measure: Number; unit: milligrams (mg) once per day
Groups:
- Part 1: All Participants (Sorafenib, Nivolumab): Participants with Child-Pugh A - B7 received a daily dose of 400mg sorafenib either once or twice a day on days 1-28, and 240mg of nivolumab IV over 30 minutes beginning on day 15 of course 1, then on days 1 and 15 of subsequent courses. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity. The course continued until 1 dose-limiting toxicity occurred to establish maximum tolerated dosing schedule.
Arm/Group | Part 1: All Participants (Sorafenib, Nivolumab)
Number analyzed (Participants) | 11
milligrams (mg) once per day | 400

2. Primary Outcome: Proportion of Participants With Grade 3 or Higher Treatment-related Adverse Events (Part 2 Only)
Description: All adverse event (AE) will be summarized based on proportion of total participants in Part 2 to evaluate the safety of the treatment combination in participants with Child-Pugh B7-9 liver function as measured by proportion of participants with an AE of toxicity grade >=3 as graded by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 and assessed as at least possibly related to sorafenib, nivolumab, or the combination of therapies.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab)
Number analyzed (Participants) | 5
proportion of participants | 0.6

3. Secondary Outcome: Proportion of Participants With Treatment-related Adverse Events
Description: Overall rates of AE and serious adverse events (SAE) as classified by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 assessed as at least possibly related to sorafenib, nivolumab, or the combination of therapies will be reported as the proportion of participants in each arm.
  .
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab)
Number analyzed (Participants) | 6 | 5 | 5
proportion of participants | 1.00 | 1.00 | 1.00

4. Secondary Outcome: Proportion of Participants Reporting Immune-related Adverse Event (irAE) (Part 1 and Part 2 Combined)
Description: Safety events for all participants assessed by treating investigator and/or Study Chair as being at least possibly immune-related while on nivolumab (irAE) will be summarized based on proportion of total participants across all treatment groups combined.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Groups:
- All Treatment Groups Combined (Sorafenib, Nivolumab): Any participants with any Child-Pugh classification who received sorafenib and nivolumab IV. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Treatment Groups Combined (Sorafenib, Nivolumab)
Number analyzed (Participants) | 16
proportion of participants | 0.94

5. Secondary Outcome: Proportion of Participants With Child-Pugh B (CPB) Reporting Immune-related Adverse Event (irAE) (Parts 1 and 2 Combined)
Description: Safety events for all CPB participants assessed by treating investigator and/or Study Chair as being at least possibly immune-related while on nivolumab (irAE) will be summarized based on proportion of total CPB participants across all treatment groups combined.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Groups:
- Parts 1 & 2: All CPB Participants: Participants with any Child-Pugh B classification across all treatment arms who received sorafenib and nivolumab IV. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Parts 1 & 2: All CPB Participants
Number analyzed (Participants) | 6
proportion of participants | 0.83

6. Secondary Outcome: Proportion of Participants With Dose Delays Due to Toxicity
Description: Delays in dosing due to adverse events will be summarized as proportion of participants by each arm.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion (Sorafenib, Nivolumab)
Number analyzed (Participants) | 6 | 5 | 5
proportion of participants | 0.833 | 1.00 | 0.8

7. Secondary Outcome: Proportion of Participants With Dose Reductions Due to Toxicity
Description: Dose reductions due to adverse events will be summarized as proportion of participants in each arm.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab)
Number analyzed (Participants) | 6 | 5 | 5
proportion of participants | 0.33 | 0.2 | 0.4

8. Secondary Outcome: Proportion of Participants Who Discontinued Treatment Due to Toxicity
Description: Treatment discontinuations due to adverse events will be summarized as proportion of participants in each arm.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab)
Number analyzed (Participants) | 6 | 5 | 5
proportion of participants | 0.167 | 0.20 | 0

9. Secondary Outcome: Proportion of Participants With an Objective Response (Part 1 and Part 2 Combined)
Description: Objective response is defined as the proportion of participants assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 with measurable disease at study entry who have an evaluated complete response (CR) or partial response (PR) at any time during the main study. Participants with measurable disease at study entry who have unknown or missing response information will be treated as non-responders.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | All Treatment Groups Combined (Sorafenib, Nivolumab)
Number analyzed (Participants) | 16
proportion of participants | 0.063

10. Secondary Outcome: Proportion of Participants With an Objective Response by Part
Description: Objective response will be based on assessments using RECIST 1.15 using local radiographic review and analyzed for Part 1 and Part 2 individually. Objective response is defined as the proportion of subjects with RECIST 1.1-measurable disease at study entry who have a CR or PR at any time during the main study. Participants with measurable disease at study entry who have unknown or missing response information will be treated as non-responders.
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Groups:
- Part 1: Combined Escalation Cohorts: Participants with Child-Pugh A-B7 who received either a daily dose of 400mg sorafenib or a twice a day dose of sorafenib on days 1-28, and 240mg of nivolumab IV over 30 minutes beginning on day 15 of course 1, then on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Part 1: Combined Escalation Cohorts | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab)
Number analyzed (Participants) | 11 | 5
proportion of participants | 0.09 | 0

11. Secondary Outcome: Median Duration of Response (DOR) (Part 1 and Part 2 Combined)
Description: DOR is defined as the median time in months from first documented evidence of complete response (CR) or partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) until the first documented sign of disease progression or death for all participant who received any treatment during the course of the study.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Treatment Groups Combined (Sorafenib, Nivolumab): All participants of any Child-Pugh classification who received sorafenib and nivolumab. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Treatment Groups Combined (Sorafenib, Nivolumab)
Number analyzed (Participants) | 16
months | 4.2 [4.2 to NA] — There were insufficient number of events so a confidence interval cannot be calculated

12. Secondary Outcome: Median Duration of Response (DOR) by Treatment Group
Description: DOR is defined as the median time in months from first documented evidence of CR or PR assessed by Response Evaluation Criteria in Solid Tumors (RECIST) until the first documented sign of disease progression or death by treatment group for all participants who received treatment during the course of the study.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part 1: Starting Dose Schedule (DL -1) Once a Day: Participants with Child-Pugh A-B7 receive a daily dose of 400mg sorafenib on days 1-28, and 240mg of nivolumab IV over 30 minutes beginning on day 15 of course 1, then on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course will continue until 1 dose-limiting toxicity occurs to establish maximum tolerated dosing schedule.
- Part 1: Escalated Dose Schedule (DL 1) Twice a Day: Participants with Child-Pugh A-B7 receive a daily dose of 400mg sorafenib twice a day on days 1-28, and 240mg of nivolumab IV over 30 minutes beginning on day 15 of course 1, then on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course will continue until 1 dose-limiting toxicity occurs to establish maximum tolerated dosing schedule.
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion (Sorafenib, Nivolumab)
Number analyzed (Participants) | 6 | 5 | 5
months | 4.2 [4.2 to NA] — There were insufficient number of events so a confidence interval could not be calculated | NA [NA to NA] — There were insufficient number of events so a confidence interval could not be calculated | NA [NA to NA] — There were insufficient number of events so a confidence interval could not be calculated

13. Secondary Outcome: Median Progression-Free Survival (PFS) (Part 1 and Part 2 Combined)
Description: PFS will be calculated as the median time in months from date of first dose of protocol therapy to date of first documented radiographic and/or clinical disease progression or death from any cause for all participants who received treatment during the course of the study. For participants who discontinued from study for other reasons than progression or death, PFS will be censored at the date last date known to be progression-free for up to 2 years following the last dose of protocol therapy.
Time Frame: Up to 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Treatment Groups Combined (Sorafenib, Nivolumab): All participants with any Child-Pugh classification who received a dose of sorafenib and nivolumab. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Treatment Groups Combined (Sorafenib, Nivolumab)
Number analyzed (Participants) | 16
months | 2.58 [2.58 to NA] — There were insufficient number of events so a confidence interval cannot be calculated.

14. Secondary Outcome: Median Progression-free Survival (PFS) by Child-Pugh Group
Description: PFS will be calculated as the median time in months from date of first dose of protocol therapy to date of first documented radiographic and/or clinical disease progression or death from any cause for participants grouped by Child-Pugh Group (Class A and Class B). For participants discontinued from study for other reasons than progression or death, PFS will be censored at the date last known to be progression-free for up to 2 years following the last dose of protocol therapy.
Time Frame: Up to 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part 1: Child-Pugh A Participants Only: Participants enrolled in Part 1 with Child-Pugh A who received at least one dose of sorafenib and nivolumab. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Parts 1 and 2: Child Pugh B Participants (Sorafenib, Nivolumab): All participants with Child-Pugh B7-9 who received at least one dose of sorafenib and nivolumab. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Part 1: Child-Pugh A Participants Only | Parts 1 and 2: Child Pugh B Participants (Sorafenib, Nivolumab)
Number analyzed (Participants) | 10 | 6
months | 2.76 [2.76 to NA] — There were insufficient number of events so a confidence interval could not be calculated | 2.58 [2.58 to NA] — There were insufficient number of events so a confidence interval could not be calculated

15. Secondary Outcome: Median Overall Survival (OS) (Part 1 and Part 2 Combined)
Description: OS is defined as the median time in months from the date of first dose of protocol therapy to the date of death due to any cause for up to 2 years following the last dose of protocol therapy. Censoring will be performed using the date of last known contact for those who are alive at the time of analysis. If data warrant, Kaplan-Meier estimates along with the 95% confidence intervals (CI) or full range will be reported.
Time Frame: Up to 3.5 years
Measure: Median (Full Range); unit: months
Arm/Group | All Treatment Groups Combined (Sorafenib, Nivolumab)
Number analyzed (Participants) | 16
months | 12.99 [1.7 to 42]

16. Secondary Outcome: Overall Survival (OS) by Child-Pugh Group
Description: OS is defined as the median time in months from the date of first dose of protocol therapy to the date of death due to any cause for up to 2 years following the last dose of protocol therapy and will be reported for each of the Child-Pugh groups separately. Censoring will be performed using the date of last known contact for those who are alive at the time of analysis. If data warrant, Kaplan-Meier estimates along with the 95% confidence intervals (CI) or full range will be reported.
Time Frame: Up to 3.5 years
Measure: Median (Full Range); unit: months
Groups:
- Part 1: Child Pugh A Participants: Participants with Child Pugh A receive sorafenib and nivolumab. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Course will continue until 1 dose-limiting toxicity occurs to establish maximum tolerated dosing schedule.
- Part 1 and 2: Child Pugh B Participants: Participants with Child Pugh B receive sorafenib and nivolumab. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Part 1: Child Pugh A Participants | Part 1 and 2: Child Pugh B Participants
Number analyzed (Participants) | 10 | 6
months | 15.26 [6.0 to 42] | 10.41 [1.7 to 36.2]

ADVERSE EVENTS:
Time Frame: Up to 3.5 years
Description: Adverse events were collected per protocol and are reported according by assigned arm regardless of any investigator directed changes to the regimen occurring after cycle 1 for Part 1 participants.
Arm/Group | Part 1: Starting Dose Schedule (DL -1) Once a Day | Part 1: Escalated Dose Schedule (DL 1) Twice a Day | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 5/6 | 2/5 | 4/5
Serious Adverse Events (participants affected / at risk) | 4/6 | 1/5 | 3/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Starting Dose Schedule (DL -1) Once a Day (N=6) | Part 1: Escalated Dose Schedule (DL 1) Twice a Day (N=5) | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab) (N=5)
Hyperbilirubinemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischemic attacks (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Starting Dose Schedule (DL -1) Once a Day (N=6) | Part 1: Escalated Dose Schedule (DL 1) Twice a Day (N=5) | Part 2: Child Pugh B Expansion Cohort (Sorafenib, Nivolumab) (N=5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 4 (10)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (2) | 2 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (6) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 3 (5) | 3 (8)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (4) | 2 (3)
Blood bilirubin increased (Investigations) | 2 (2) | 3 (6) | 2 (2)
Weight loss (Investigations) | 3 (3) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (6) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (4) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 0 (0) | 3 (3)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The Part 2 Child Pugh B Expansion Cohort was closed to further accrual earlier than expected due to slow accrual resulting from a changing treatment landscape in hepatocellular carcinoma (HCC) with multiple new drug approvals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT03439891/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT03439891/ICF_001.pdf